CLINICAL TRIAL: NCT00006332
Title: Treatment of Hepatocellular Carcinoma With Tetrathiomolybdate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: NCRR-M01RR00042-1707; M01RR000042 (NIH)
Record Dates: First submitted 2000-10-04; First posted 2000-10-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Molybdenum
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tetrathiomolybdate

INTERVENTIONS:
Drug: Tetrathiomolybdate

SUMMARY:
Hepatocellular carcinoma (HCC) is a deadly tumor for which the incidence is increasing in the United States, primarily due to prevalence of hepatitis C infection. An important aspect of the development of HCC is that it occurs in patients who have underlying cirrhosis of the liver, thereby limiting the therapeutic options. There is potential curative treatment for these patients, such as resection of the tumor lesion and liver transplantation, but these treatments are feasible in a small percent of patients only. Furthermore, the majority of the patients with HCC are also not candidates for palliative treatments such as percutaneous ablation of the tumor, chemotherapy or radiation. Additionally, it has been shown that these palliative treatment modalities do not alter survival, and are associated with significant risks. Therefore, there are no treatment options for most patients with HCC. A new theory has emerged in the fight against cancer through inhibition of angiogenesis (development of new blood vessels). The hypothesis being that if there is no blood supply "feeding" the tumor cells cannot divide or survive. One such approach, pioneered in this institution by Drs. George Brewer and Sofia Merajver, is the anticopper approach using the medication tetrathiomolybdate (TM). By creating a mild copper deficiency state, several pathways required for angiogenesis are inhibited. They performed a Phase I trial in which patients with metastatic cancer were treated with TM resulting in decrease tumor vascularity. TM had excellent safety profile in this patient population. HCC is well known to be a hypervascular tumor. An antiangiogenesis approach might provide a novel treatment for this HCC. This is a pilot study of 10 patients with HCC who are not candidates for curative surgical therapy with resection or liver transplantation, nor for ablative techniques. Patients seen in the General Liver clinic and Liver Transplant clinic who have an overall good performance status, with an expected survival of more than 6 months will be enrolled. After an initial evaluation, they will be given 120 mg/day of TM in divided doses for one year. The size and vascularity of the tumor will be evaluated by magnetic resonance imaging (MRI). The primary outcome of this study is to prevent tumor progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with definite diagnosis of HCC based on a Dynamic MRI revealing a vascular mass in the liver and histologic confirmation of HCC.
* Patients who are not candidates for surgical resection, OLT or radiofrequency ablation.
* Patients with no prior treatment for HCC.
* Patients with extrahepatic spread and/or vascular invasion are permissible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- 3912 Taubman Center, Ann Arbor, Michigan, United States